CLINICAL TRIAL: NCT01343043
Title: A Pilot Study of Genetically Engineered NY-ESO-1 Specific NY-ESO-1ᶜ²⁵⁹T in HLA-A2+ Patients With Synovial Sarcoma
Acronym: NY-ESO-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 208466; ADP 04511 (Other: Adaptimmune Therapeutics); 2015-005594-21 (EudraCT Number)
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Neoplasms
Keywords: T Cell Receptor; Sarcoma; Cell Therapy; T Cell Therapy; Previously treated; NY-ESO-1; Metastatic; Immuno-oncology
MeSH Terms: conditions — Neoplasms; Sarcoma; Neoplasm Metastasis | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Cohort 1 treated with NY-ESO-1 T Cells (Experimental): High NY-ESO-1 expression and the use of cyclophosphamide plus fludarabine as the lymphodepleting chemotherapy.
  Interventions: Drug: NY-ESO-1(c259)T Cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Cohort 2 treated with NY-ESO-1 T Cells (Experimental): Low NY-ESO-1 expression and the use of cyclophosphamide plus fludarabine as the lymphodepleting chemotherapy.
  Interventions: Drug: NY-ESO-1(c259)T Cells; Drug: Fludarabine; Drug: Cyclophosphamide
- Cohort 3 treated with NY-ESO-1 T Cells (Experimental): High NYESO-1 expression and the use of cyclophosphamide only for lymphodepletion rather than fludarabine as the lymphodepleting chemotherapy.
  Interventions: Drug: NY-ESO-1(c259)T Cells; Drug: Cyclophosphamide
- Cohort 4 treated with NY-ESO-1 T Cells (Experimental): High NY-ESO-1 expression and the use of reduced dose cyclophosphamide plus fludarabine regimen as the lymphodepleting chemotherapy.
  Interventions: Drug: NY-ESO-1(c259)T Cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: NY-ESO-1(c259)T Cells — Lymphodepleting chemotherapy followed by infusion with NY-ESO-1(c259) transduced autologous T cells. Subjects will receive one infusion of NY-ESO-1 genetically engineered T cells on Day 0.
Drug: Fludarabine — Fludarabine will be used as lymphodepleting chemotherapy.
  Arms: Cohort 1 treated with NY-ESO-1 T Cells; Cohort 2 treated with NY-ESO-1 T Cells; Cohort 4 treated with NY-ESO-1 T Cells
Drug: Cyclophosphamide — Cyclophosphamide will be used as lymphodepleting chemotherapy.

SUMMARY:
The purpose of this early (pilot) clinical trial is to test the effects (both good and bad) of chemotherapy and adoptive immunotherapy with T cells engineered to recognize NY-ESO-1 peptide in patients with unresectable, metastatic or recurrent synovial sarcoma.

DETAILED DESCRIPTION:
Design

* Patients will undergo apheresis at the enrolling institution. PBMC will be shipped to a central manufacturer for gene transduction, activation and expansion, then cryopreserved and shipped back to the enrolling institution.
* The trial seeks to enroll up to 65 patients, that is, up to 20 patients in Cohort 1 and up to 15 patients in Cohorts 2-4. Depending on the cohort patients are enrolled in, patients will undergo lymphodepletion with cyclophosphamide with or without fludarabine.

  * Cohort 1: Complete
  * Cohort 2: Up to 15 patients may be enrolled to achieve at least 10 evaluable patients treated with NY-ESO-1ᶜ²⁵⁹T. Patients will undergo lymphodepletion with cyclophosphamide plus fludarabine on Days -3 and -2, and without fludarabine on Days -5 and -4.
  * Cohort 3: Up to 15 patients may be enrolled to achieve at least 10 evaluable patients treated with NY-ESO-1ᶜ²⁵⁹T. Patients will undergo lymphodepletion with cyclophosphamide only on Days -3 and -2. (Cohort Complete)
  * Cohort 4: Up to 15 patients may be enrolled to achieve at least 5 evaluable patients treated with NY-ESO-1ᶜ²⁵⁹T. Patients will undergo lymphodepletion with cyclophosphamide plus fludarabine on Days -7 to -5.

On Day 0, patients ≥40 kg will receive the minimum cell dose of at least 1x10⁹ transduced NY-ESO-1ᶜ²⁵⁹T cells with a maximum of 6x10⁹ transduced cells. The target dose for this protocol is 5x10⁹ transduced NY-ESO-1ᶜ²⁵⁹T cells. Patients <40 kg will be dosed per body weight with a minimum 0.025x10⁹ transduced cells/kg, with a target dose of 0.125 x10⁹ transduced cells/kg.

* Patients will be monitored for toxicity, antitumor effects and immune endpoints.
* Patients who have a confirmed response, or have stable disease for >3 months then progress may receive a 2nd T cell infusion, provided eligibility criteria are met. The 2nd treatment cell infusion will be administered in the same manner as the first. Patients who meet the eligibility criteria may receive a 2nd infusion of NY-ESO-1ᶜ²⁵⁹T no sooner than 60 days and no later than 2 years following completion of the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Synovial sarcoma that has been treated with standard chemotherapy containing ifosfamide and/or doxorubicin and remains: unresectable or metastatic or progressive/persistent or recurrent disease
* Measurable disease
* Patients must have proven positive tumor sample for NY-ESO-1 as follows:

  * Cohort 1 -Positive expression is defined as 2+ and/or 3+ by immunohistochemistry in ≥ 50% of cells.
  * Cohort 2 -Positive expression is defined as ≥1+ by immunohistochemistry in ≥1% cells, but not to exceed 2+ and/or 3+ in ≥ 50% of cells.
  * Cohort 3 -Positive expression is defined as 2+ and/or 3+ by immunohistochemistry in ≥ 50% of cells.
  * Cohort 4 -Positive expression is defined as 2+ and/or 3+ by immunohistochemistry in ≥ 50% of cells.
* HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 by high resolution testing at a local or central laboratory
* Weigh more than 18 kg
* All previous cytotoxic chemotherapy, monoclonal antibody therapy, or immune therapy must be washed out 3 weeks before apheresis and must be completed at least 3 weeks prior to pre-infusion lymphodepletive chemotherapy.
* Systemic corticosteroid or other immunosuppressive therapy should be washed out 2 weeks before apheresis and must be completed at least 2 weeks prior to pre-infusion lymphodepletive chemotherapy.
* Biologic or other approved molecular targeted small molecule inhibitors should be washed out 1 week or 5 half-lives (whichever is longer) before apheresis and must be completed at least 1 week or 5 half-lives (whichever is longer) prior to pre-infusion lymphodepletive chemotherapy.
* Any grade 3 or 4 hematologic toxicity of any previous therapy must have resolved to grade 2 or less prior to apheresis and any grade 3 or 4 toxicity must have resolved to grade 2 or less prior to pre-infusion lymphodepletive chemotherapy.
* ECOG 0-1, or for children ≤10 years of age, Lansky > 60
* Life expectancy > 3 months
* Left ventricular ejection fraction ≥ 40% or fractional shortening ≥ 28%
* T. bilirubin < 2 mg/dl (Patients with Gilbert Syndrome total bilirubin <3xULN and direct bilirubin ≤ 35%)
* AST, ALT ≤ 2.5 x upper limit of normal
* ANC ≥ 1.0 x 10⁹/L
* Platelets ≥ 75 x 10⁹/L
* Age-adjusted normal serum creatinine or a creatinine clearance ≥ 40 ml/min
* Ability to give informed consent for patients greater than 18 years of age. For patients less than 18 years of age the legal guardian must give informed consent.
* Male patients must be willing to practice birth control (including abstinence) during and for 4 months after treatment. Female patients must be willing to practice birth control (including abstinence) during treatment and for 4 months after gene modified cells are no longer detected in body.

Exclusion Criteria:

* Active HIV, HBV, HCV or HTLV 1/2 infection (due to increased risk of complications during lymphodepleting regimen and confounding effects on the immune system). Active hepatitis B or C infection is defined by seropositive for hepatitis B surface antigen (HbSAg) or hepatitis C antibody.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Investigational Site, Duarte, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Houston, Texas

REFERENCES:
- [Derived] Gyurdieva A, Zajic S, Chang YF, Houseman EA, Zhong S, Kim J, Nathenson M, Faitg T, Woessner M, Turner DC, Hasan AN, Glod J, Kaplan RN, D'Angelo SP, Araujo DM, Chow WA, Druta M, Demetri GD, Van Tine BA, Grupp SA, Fine GD, Eleftheriadou I. Biomarker correlates with response to NY-ESO-1 TCR T cells in patients with synovial sarcoma. Nat Commun. 2022 Sep 8;13(1):5296. doi: 10.1038/s41467-022-32491-x. PMID 36075914
- [Derived] Ramachandran I, Lowther DE, Dryer-Minnerly R, Wang R, Fayngerts S, Nunez D, Betts G, Bath N, Tipping AJ, Melchiori L, Navenot JM, Glod J, Mackall CL, D'Angelo SP, Araujo DM, Chow WA, Demetri GD, Druta M, Van Tine BA, Grupp SA, Abdul Razak AR, Wilky B, Iyengar M, Trivedi T, Winkle EV, Chagin K, Amado R, Binder GK, Basu S. Systemic and local immunity following adoptive transfer of NY-ESO-1 SPEAR T cells in synovial sarcoma. J Immunother Cancer. 2019 Oct 24;7(1):276. doi: 10.1186/s40425-019-0762-2. PMID 31651363
- [Derived] D'Angelo SP, Melchiori L, Merchant MS, Bernstein D, Glod J, Kaplan R, Grupp S, Tap WD, Chagin K, Binder GK, Basu S, Lowther DE, Wang R, Bath N, Tipping A, Betts G, Ramachandran I, Navenot JM, Zhang H, Wells DK, Van Winkle E, Kari G, Trivedi T, Holdich T, Pandite L, Amado R, Mackall CL. Antitumor Activity Associated with Prolonged Persistence of Adoptively Transferred NY-ESO-1 c259T Cells in Synovial Sarcoma. Cancer Discov. 2018 Aug;8(8):944-957. doi: 10.1158/2159-8290.CD-17-1417. Epub 2018 Jun 11. PMID 29891538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was designed to determine whether New York esophageal squamous cell carcinoma 1 (NY-ESO-1) specific genetically engineered T cells recognized a human leukocyte antigens (HLA-A2) binding peptide from NY-ESO-1 induced antitumor responses in participants with synovial sarcoma.
Pre-assignment Details: A total of 50 participants were enrolled in this study. Out of 50 participants, 45 participants received NY-ESO-1 genetically engineered T cell infusion.
Groups:
- Cohort 1: High NY-ESO-1 Expression Treated With Regimen A: Participants with high tumor expression of NY-ESO-1 underwent lymphodepletion with regimen A (lymphodepleting chemotherapeutic agents; cyclophosphamide plus fludarabine on Days -3 and -2, intravenously [IV] and only fludarabine on Days -5 and -4, IV). Participants received one infusion of NY-ESO-1 genetically engineered T cells on Day 0. High tumor NY-ESO-1 expression was defined as 2+ or 3+ by immunohistochemistry (IHC) in >=50% cells.
- Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A: Participants with low tumor expression of NY-ESO-1 underwent lymphodepletion with regimen A (lymphodepleting chemotherapeutic agents; cyclophosphamide plus fludarabine on Days -3 and -2, IV and only fludarabine on Days -5 and -4, IV). Participants received one infusion of NY-ESO-1 genetically engineered T cells on Day 0. Low tumor NY-ESO-1 expression was defined as >=1+ by IHC in >=1% cells but not to exceed 2+ or 3+ in >=50% cells..
- Cohort 3: High NY-ESO-1 Expression Treated With Regimen B: Participants with high tumor expression of NY-ESO-1 underwent lymphodepletion with regimen B (lymphodepleting chemotherapeutic agent; cyclophosphamide only on Days -3 and -2, IV). Participants received one infusion of NY-ESO-1 genetically engineered T cells on Day 0. High tumor NY-ESO-1 expression was defined as 2+ or 3+ by immunohistochemistry (IHC) in >=50% cells.
- Cohort 4: High NY-ESO-1 Expression Treated With Regimen C: Participants with high tumor expression of NY-ESO-1 underwent lymphodepletion with regimen C (lymphodepleting chemotherapeutic agents; reduced dose of cyclophosphamide plus fludarabine on Days -7 to -5, IV). Participants received one infusion of NY-ESO-1 genetically engineered T cells on Day 0. High tumor NY-ESO-1 expression was defined as 2+ or 3+ by immunohistochemistry (IHC) in >=50% cells.
Period: Overall Study
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Started | 15 | 14 | 5 | 16
Received T-cell Infusion | 12 | 13 | 5 | 15
Completed | 12 | 13 | 5 | 15
Not Completed | 3 | 1 | 0 | 1
Not completed — Disease progression before treatment | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C | Total
Number analyzed (Participants) | 15 | 14 | 5 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.5 (10.00) | 33.1 (16.18) | 25.4 (8.73) | 41.2 (13.80) | 33.6 (14.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 2 | 8 | 25
  Male | 7 | 7 | 3 | 8 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 13 | 11 | 4 | 15 | 43
  Missing | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was calculated as the percentage of participants with a confirmed complete response (CR) or partial response (PR) relative to the total number of participants in the analysis population per response evaluation criteria in solid tumors (RECIST) version (v)1.1 as determined by the local investigators.
Time Frame: Up to 4.5 years
Population: Modified intent-to-treat (mITT) Population comprised of all participants who received NY-ESO-1 genetically engineered T cell infusion
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 12 | 13 | 5 | 15
Percentage of Participants | 50 | 30.8 | 20 | 26.7

2. Secondary Outcome: Duration of Overall Response
Description: Duration of overall response (DOR) is defined as the time from first documented evidence of confirmed CR or confirmed PR until first documented date of disease progression or death due to any cause or surgical resection or start of prohibited medications. Duration of overall response was evaluated per RECIST v1.1. Median and full range of DOR are presented.
Time Frame: Up to 4.5 years
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 6 | 4 | 1 | 4
Weeks | 31.0 [13 to 72] | 8.6 [8 to 13] | 32.1 [NA to NA] — Full range is not applicable due to single participant, and the median value presented here is the actual DOR for this single participant. | 16.4 [14 to 94]

3. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the interval between the date of first T cell infusion and the earliest documented evidence of disease progression or death due to any cause or surgical resection or start of prohibited medications. Progression free survival was evaluated per RECIST v1.1. Median and inter-quartile range (first quartile and third quartile) of progression free survival are presented.
Time Frame: Up to 4.5 years
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 12 | 13 | 5 | 15
Weeks | 15.4 [8.6 to 37.1] | 13.1 [8.3 to 13.9] | 8.6 [8.3 to 12.1] | 22.4 [11.6 to 38.3]

4. Secondary Outcome: Best Overall Response
Description: Best overall response is the best response recorded from the start of treatment (first T cell infusion) until disease progression/recurrence. Response categories from best to worst are confirmed CR, confirmed PR, stable disease (SD) and confirmed progressive disease (PD). Best overall response is a stable disease, if CR or PR are unconfirmed. Data for number of participants with CR, PR, SD and PD are presented.
Time Frame: Up to 4.5 years
Population: mITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 12 | 13 | 5 | 15
Participants
  Complete response | 1 | 0 | 0 | 0
  Partial response | 5 | 4 | 1 | 4
  Stable disease | 5 | 7 | 3 | 10
  Progressive disease | 1 | 1 | 0 | 1
  Not evaluable | 0 | 1 | 1 | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the interval between the date of the first T-cell infusion and date of death from any cause. Median and inter-quartile range (first quartile and third quartile) of overall survival are presented.
Time Frame: Up to 4.5 years
Population: mITT Population
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 12 | 13 | 5 | 15
Weeks | 80.7 [45.3 to 212.0] | 43.1 [19.4 to 85.3] | 86.4 [68.1 to 104.6] | 105.3 [50.3 to NA] — <75% of participants experienced the event within the treatment arm. Hence, third quartile could not be derived.

6. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations judged by physician, is associated with liver injury and impaired liver function. Number of participants who had non-SAEs and SAEs are presented.
Time Frame: Up to 5 years
Population: Intent-to-treat (ITT) Population comprised of all participants who were enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 15 | 14 | 5 | 16
Participants
  Non-SAE | 15 | 13 | 5 | 15
  SAE | 9 | 7 | 4 | 6

7. Secondary Outcome: Number of Participants With Worst Post-Baseline Grade Results for Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters. No data collected separately for this outcome measure as any abnormal value would be recorded as an adverse event.
Time Frame: Up to 4.5 years
Population: mITT Population
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Worst Post-Baseline Grade Results for Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters. No data collected separately for this outcome measure as any abnormal value would be recorded as an adverse event.
Time Frame: Up to 4.5 years
Population: mITT Population
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-Baseline Anti-infused (NY-ESO-1 Genetically Engineered T) Cell Antibody Result
Description: Serum samples were collected for the determination of anti-infused (NY-ESO-1 genetically engineered T) cell antibodies (ATA) using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. A participant was considered to have a confirmed positive ATA result if they have a positive screening assay result and a positive confirmation assay result.
Time Frame: Up to 4.5 years
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 10 | 8 | 3 | 8
Participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Concentration of Cytokines in Cytokine Release Syndrome (CRS) by CRS Status: Cohort 1: High NY-ESO-1 Expression Treated With Regimen A
Description: CRS is a potentially life-threatening toxicity that is observed following administration of antibodies and adoptive T-cell therapies for cancer. Serum samples were collected to analyze the concentration of cytokines using the electrochemiluminescent tagged detection antibodies. The correlation between cytokines and cytokine release syndrome was considered between participants who had serious CRS vs no CRS or Non-serious CRS. There were only 4 participants across the whole study that had serious CRS and cytokine data was available for 3 of these participants. Due to the limited number of participants that had serious CRS no statistical correlations in cytokine levels and CRS could be performed. A listing of the levels of cytokines for the 3 participants with serious CRS is available/provided.
Time Frame: Up to Week 4
Population: mITT Population.
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A
Number analyzed (Participants) | 0

11. Secondary Outcome: Concentration of Cytokines in CRS by CRS Status: Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A
Description: as for outcome 10
Time Frame: Up to Week 4
Population: mITT Population.
Arm/Group | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A
Number analyzed (Participants) | 0

12. Secondary Outcome: Concentration of Cytokines in CRS by CRS Status: Cohort 3: High NY-ESO-1 Expression Treated With Regimen B
Description: as for outcome 10
Time Frame: Up to Week 4
Population: mITT Population
Arm/Group | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B
Number analyzed (Participants) | 0

13. Secondary Outcome: Concentration of Cytokines in CRS by CRS Status: Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Description: as for outcome 10
Time Frame: Up to Week 4
Population: mITT Population.
Arm/Group | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0

14. Secondary Outcome: Time to Maximum Persistence of NY-ESO-1 Genetically Engineered T Cells
Description: Time to maximum persistence is defined as date of maximum persistence for infusion visit minus date of first T cell infusion visit plus 1. Median and full range of time to maximum persistence are presented.
Time Frame: Up to 4.5 years
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Days
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 6 | 4 | 1 | 4
Days | 8.0 [4 to 29] | 8.0 [5 to 18] | 8.0 [8 to 8] | 9 [6 to 13]

15. Other Pre Specified Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was planned to be evaluated. An event was to be considered a DLT if it occurred within the first 21 days of treatment, and met one of the protocol defined DLT criteria. The results for this outcome measure will never be posted.
Time Frame: Up to Day 21 (from first dose)
Population: mITT Population. This was an other pre-specified outcome measure. The results for this outcome measure will never be posted.
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Other Pre Specified Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram, Echocardiogram and Multigated Acquisition Scan Findings
Description: Abnormal electrocardiogram, echocardiogram and multigated acquisition scan findings were planned to be evaluated. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee. The results for this outcome measure will never be posted.
Time Frame: Up to 4.5 years
Population: as for outcome 15
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Other Pre Specified Outcome: Percentage of Participants With Confirmed CR
Description: Participants were planned to be evaluated for confirmed CR according to RECIST v1.1, after receiving a second dose of NY-ESO-1 genetically engineered T cell infusion. The results for this outcome measure will never be posted.
Time Frame: Up to 4.5 years
Population: as for outcome 15
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment (Day 1) until maximum of 4.5 years
Description: SAEs and non-serious AEs were reported for the ITT Population which comprised of all participants who were enrolled in the study.
Arm/Group | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C
All-Cause Mortality (participants affected / at risk) | 12/15 | 13/14 | 4/5 | 8/16
Serious Adverse Events (participants affected / at risk) | 9/15 | 7/14 | 4/5 | 6/16
Other Adverse Events (participants affected / at risk) | 15/15 | 13/14 | 5/5 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A (N=15) | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A (N=14) | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B (N=5) | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C (N=16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 0 | 3
Chills (General disorders) | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 2 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 3 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: High NY-ESO-1 Expression Treated With Regimen A (N=15) | Cohort 2: Low NY-ESO-1 Expression Treated With Regimen A (N=14) | Cohort 3: High NY-ESO-1 Expression Treated With Regimen B (N=5) | Cohort 4: High NY-ESO-1 Expression Treated With Regimen C (N=16)
Fatigue (General disorders) | 12 | 8 | 3 | 14
Pyrexia (General disorders) | 12 | 10 | 4 | 9
Oedema peripheral (General disorders) | 4 | 5 | 1 | 3
Pain (General disorders) | 3 | 2 | 2 | 6
Chills (General disorders) | 2 | 3 | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 4 | 3 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 4
Asthenia (General disorders) | 0 | 1 | 0 | 3
Injection site reaction (General disorders) | 2 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 2
Malaise (General disorders) | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0 | 1
Tenderness (General disorders) | 1 | 1 | 0 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0 | 0
Catheter site irritation (General disorders) | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1
Catheter site vesicles (General disorders) | 0 | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 12 | 10 | 5 | 12
Lymphocyte count decreased (Investigations) | 13 | 8 | 3 | 7
Neutrophil count decreased (Investigations) | 11 | 8 | 4 | 7
Platelet count decreased (Investigations) | 12 | 7 | 4 | 7
Alanine aminotransferase increased (Investigations) | 6 | 4 | 3 | 4
Blood creatinine increased (Investigations) | 8 | 2 | 1 | 4
Activated partial thromboplastin time prolonged (Investigations) | 9 | 3 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 7 | 4 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 7 | 1 | 2 | 2
Weight decreased (Investigations) | 2 | 4 | 2 | 2
Lipase increased (Investigations) | 6 | 0 | 0 | 0
Amylase increased (Investigations) | 2 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 2 | 1
Breath sounds abnormal (Investigations) | 0 | 2 | 1 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 2 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 2 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 2 | 0 | 0 | 0
Serum ferritin increased (Investigations) | 0 | 1 | 1 | 0
Urine output decreased (Investigations) | 1 | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 1
Cytomegalovirus test positive (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 0 | 0 | 1
Epstein-Barr virus antibody positive (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 14 | 13 | 4 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 4 | 0 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 13 | 10 | 4 | 13
Diarrhoea (Gastrointestinal disorders) | 8 | 9 | 2 | 5
Vomiting (Gastrointestinal disorders) | 7 | 6 | 3 | 6
Constipation (Gastrointestinal disorders) | 8 | 3 | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Proctalgia (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Scalloped tongue (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 7 | 3 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 7 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 5 | 5 | 2 | 7
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 4 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 6 | 1 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 4 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 1 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1
Appetite disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 2 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 2 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 7 | 7 | 2 | 4
Tachycardia (Cardiac disorders) | 4 | 4 | 2 | 6
Pericardial effusion (Cardiac disorders) | 1 | 0 | 2 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Pulmonary valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 4 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 3 | 3 | 4
Headache (Nervous system disorders) | 8 | 1 | 3 | 7
Paraesthesia (Nervous system disorders) | 4 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 2 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 2 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Phantom limb syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 10 | 3 | 0 | 6
Insomnia (Psychiatric disorders) | 4 | 5 | 0 | 3
Depression (Psychiatric disorders) | 3 | 1 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 3 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 2 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Social avoidant behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 4 | 8 | 2 | 7
Hypertension (Vascular disorders) | 2 | 3 | 2 | 5
Hot flush (Vascular disorders) | 3 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 1 | 0
Flushing (Vascular disorders) | 1 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 1 | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 1 | 0 | 0 | 0
Groin infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 4 | 5 | 3 | 4
Hypersensitivity (Immune system disorders) | 0 | 3 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 2 | 2 | 1
Haematuria (Renal and urinary disorders) | 1 | 3 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0
Fanconi syndrome acquired (Renal and urinary disorders) | 1 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 2
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 2
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Premature menopause (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pruritus genital (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT01343043/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01343043/SAP_001.pdf